

## Association of Hepatitis C Virus With Breast Cancer

NCT04090164



MAY 20, 2020
© Osama Hussein
Mansoura University

## Participants flow chart



The Hospital records were searched for "malignant neoplasm of the breast" diagnosis. All consecutive patients treated at the surgery department from January 2013 through December 2018 were identified. The list of identified patients was alphabetically arranged and the data of an unselected sample of those patients was retrieved from the system.

The following information were collected for all patients: name, age, hospital number, tumor stage information (T,N,M), tumor grade, tumor biological type, anti-HCV serological status at diagnosis, Hepatitis B surface antigen status at diagnosis and the date and status at the last hospital visit.

Mann-Whitney, Chi-square and Log-rank tests were used for comparison of anti-HCV positive with anti-HCV negative patients regarding age, tumor characteristics and disease-free survival (DFS) respectively.

The data from a published population-based study was used as a measurement of anti-HCV status in the non-cancer adult female population of Dakahlia [1] and (El-Ghitany; unpublished communication). Fisher's exact test was used to compare the proportions of seropositive cases in the breast cancer cohort to that of the Dakahlia population.

Statistical calculations used GraphPad Quick Calculator and GraphPad Prism© V.4 (GraphPad Software, Inc.).

1. El-Ghitany EM, Farghaly AG (2019) Geospatial epidemiology of hepatitis C infection in Egypt 2017 by governorate. Heliyon 5 (8):e02249. doi:10.1016/j.heliyon.2019.e02249